CLINICAL TRIAL: NCT05880979
Title: Engaging Together for Healthy Relationships: A Pilot Trial to Test a Brief Dating Violence Prevention Intervention for Pediatric Primary Care
Brief Title: Engaging Together for Healthy Relationships
Acronym: ETHR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Maya Ragavan, Assistant Professor of Pediatrics, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY22060047
Record Dates: First submitted 2023-05-12; First posted 2023-05-30 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Violence in Adolescence; Domestic Violence

STUDY DESIGN:
Intervention Model Description: Randomization will occur at the provider-level
Who Masked: Participant
Masking Description: Participants will be told in the consent form that they may receive information about dating violence during their well-visit or they may not. They will not be specifically told if their provider is the intervention provider or control provider.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Engaging Together for Healthy Relationships) (Experimental): Providers and families in the intervention arm will receive the ETHR program which includes a clinician training, provider scripts, resource guides, a comprehensive website, and warm referral processes.
  Interventions: Behavioral: Engaging Together for Healthy Relationships
- Control (Receipt of regular well-child care) (Active Comparator): Providers and families in the control arm will receive regular well-child care. All providers in the control arm will have access to ETHR after the pilot trial is over
  Interventions: Behavioral: Regular well child care

INTERVENTIONS:
Behavioral: Engaging Together for Healthy Relationships — A comprehensive parent-adolescent dating violence prevention intervention designed to be provider delivered within the context of a pediatric well-child visit
  Arms: Intervention (Engaging Together for Healthy Relationships)
Behavioral: Regular well child care — Participants will receive their regularly scheduled well-child care
  Arms: Control (Receipt of regular well-child care)

SUMMARY:
The goal of this pilot randomized clinical trial is to assess feasibility and acceptability of a brief parent-adolescent dating violence prevention intervention (Engaging Together for Healthy Relationships; ETHR) delivered in pediatric primary care settings. The main questions it aims to answer is if ETHR is acceptable and feasible. 4 healthcare providers will receive ETHR to share with their patients which includes clinician training, provider-delivered scripts, resource guides, and a comprehensive website. This will be compared to providers conducting routine well-child care with their patients.

DETAILED DESCRIPTION:
The investigators are conducting a pilot randomized clinical trial to test a brief parent-adolescent dating violence prevention intervention (Engaging Together for Healthy Relationships; ETHR). ETHR has been developed for parents and adolescents, to be implemented within pediatric primary care settings. ETHR is a comprehensive intervention which includes a training for clinicians, brief educational scripts for providers, resource guides for the adolescent, parent, and dyad, a comprehensive website, and warm referral processes to connect families with local resources. The investigators will be comparing ETHR with routine care. The specific goal of the pilot trial is to test trial feasibility, as well as intervention acceptability and fidelity. The investigators also will be examining exploratory changes in secondary outcomes and early implementation barriers and facilitators.

Four pediatric clinics will participate in this study. The investigator will recruit two providers from each clinic and randomize them into the intervention provider or control provider. The intervention provider will receive ETHR and the control provider will complete their regular well-child care. The investigators will enroll 15 families in the intervention arm and 5 in the control arm (3:1 enrollment). Families who are seeing the intervention provider for a well-child visit will be enrolled in the intervention arm; those seeing the control provider will be enrolled in the control arm. Families will be eligible if they are seeing the intervention or control providers for a well child visit, if the adolescent coming for the well-visit is between 11 to 15, if both the caregiver and adolescent are interested in participating, and if the family speaks and understands English. Families will be called 2 weeks ahead of their visit to enroll, consent, and complete a baseline survey (both the adolescent and parent will complete the survey). Participants will then attend their well -visit (where they will receive ETHR or routine care, depending on their provider). They will complete an acceptability and fidelity survey immediately post-visit, a resource utilization survey 1 month post visit, and a follow up survey (identical to the baseline survey) 3 months post visit. Providers will complete a brief fidelity and acceptability survey after each study visit (15 for intervention providers, 5 for control providers). All providers and a subset of families enrolled in the intervention arm (20 dyads, 40 participants) will also complete post-intervention interviews.

ELIGIBILITY:
Inclusion Criteria:

Providers:

1. Sees patient at an eligible primary care clinic
2. Speaks and understands English
3. Age 18 or older
4. Identifies as a pediatrician, nurse practitioner, physician assistant (pediatric primary care healthcare provider)

Adolescents

1. Age 11 to 15
2. Attending an upcoming well-child visit from a provider enrolled in the study
3. Caregiver who is accompanying well-child visit with adolescent is also participating
4. Speaks and understands English

Parents

1. Is parent or primary caregiver for an adolescent age 11 to 15
2. Adolescent has an upcoming well-child visit with a provider enrolled in the study
3. Accompanying child to the well-visit
4. Adolescent is interested and eligible to participate in study
5. Speaks and understand English

Exclusion Criteria:

Providers

1) Does not need inclusion criteria

Min Age: 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Percentage of participants who are eligible out of the total who are approached | Through completion of study recruitment, an average of 6 months
  Will assess through tracking data
Percentage of participants who are consented out of the total who are eligible | Through completion of study recruitment, an average of 6 months
  Will assess through tracking data
Percentage of participants who complete the baseline survey out of the total who consented | Through completion of completing baseline surveys, an average of 6 months
  Will assess through tracking data
Percentage of participants who complete the well-visit out of the total who consented | Through completion of completing well-visits, an average of 6 months
  Will assess through tracking data
Percentage of participants who complete the immediate post-intervention survey out of the total who consented | Through completion of completing post-intervention survey, an average of 7 months
  Will assess through tracking data
Percentage of participants who complete the 1-month post-intervention survey out of the total who consented | 4 months
  Through completion of completing 1- month post-intervention survey, an average of 8 months
Percentage of participants who complete the 3-month post-intervention survey out of the total who consented | Through completion of completing 3 month post-intervention survey, an average of 12 months
  Will assess through tracking data
Percentage of participants who strongly agree or agree that the intervention is acceptable using a 4-item validated measure (Acceptability of Intervention Measure) | Through completion of completing immediate post-visit surveys, an average of 6 months
  Validated measure (Acceptability of Intervention Measure)

SECONDARY OUTCOMES:
Self-efficacy in preventing adolescent relationship abuse (ARA), change in outcome between baseline and 3 months | Baseline, 3-month post intervention
  Self-efficacy around ARA prevention, 1-5 scale (5=higher self-efficacy)
Percentage of participants who utilize ARA resources at each measurement point, change in outcome over time | Baseline, 1 month post intervention, 3 month post-intervention
  Investigator developed measure (yes/no)
Attitudes about ARA, change in outcome between baseline and 3 months | Baseline, 3-month post intervention
  Attitudes about Abusive Relationships, 1-5 scale (1=not abusive, 5=very abusive)
Parent-adolescent communication around dating and ARA, change in outcome over time | Baseline, 3-month post intervention
  Investigator developed measure, yes/no answer choices (yes=has communicated, no=has not communicated)
Parental monitoring around dating and ARA, change in outcome over time | Baseline, 3-month post intervention
  Parenting Practices Scale (never to always; 1=never, 5=always)
Percentage of adolescents reporting ARA victimization and perpetration | Baseline, 3-month post intervention
  CADRI Short Form 1-5 scale (never to everyday)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - CCP South Hills, Monongahela, Pennsylvania
  - Primary Care Center Oakland, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided